CLINICAL TRIAL: NCT01817166
Title: Multicentric, Randomized, Double-blind Versus Placebo Study Evaluating the Efficacy of Treatment With Cholecalciferol (Vitamin D3) for Delaying the Diagnosis of Multiple Sclerosis (MS) After a Clinically Isolated Syndrome (CIS). Comparison of Conversion Rates After 2 Years.
Brief Title: Efficacy of Cholecalciferol (Vitamin D3) for Delaying the Diagnosis of MS After a Clinically Isolated Syndrome
Acronym: D-Lay-MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PHRC-N/2012/ET-01; 2012-005821-59 (EudraCT Number)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: cholecalciferol; vitamin D; immune disease; clinically isolated syndrome
MeSH Terms: conditions — Multiple Sclerosis; Immune System Diseases | interventions — Vitamin D; Cholecalciferol; X-Rays; Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients in this arm will receive a placebo treatment mimicking 100.000 UI of cholecalciferol every 14 days for a maximum of 24 months or until conversion to full multiple sclerosis has occurred.
  Intervention: Placebo Intervention: Imaging Intervention: Lumbar puncture Intervention: Blood sampling Intervention: Urine samples
  Interventions: Drug: Placebo; Other: Imaging; Biological: Lumbar puncture; Biological: Blood sampling; Biological: Urine samples
- Vit D (Experimental): Patients in this arm will receive 100.000 UI of cholecalciferol every 14 days for a maximum of 24 months or until conversion to full multiple sclerosis has occurred.
  Intervention: Vitamin D Intervention: Imaging Intervention: Lumbar puncture Intervention: Blood sampling Intervention: Urine samples
  Interventions: Drug: Vitamin D; Other: Imaging; Biological: Lumbar puncture; Biological: Blood sampling; Biological: Urine samples

INTERVENTIONS:
Drug: Vitamin D — Patients will receive 100.000 UI of cholecalciferol every 14 days for a maximum of 24 months or until conversion to full multiple sclerosis has occurred.
  Other Names: Cholecalciferol
  Arms: Vit D
Drug: Placebo — Patients will receive a placebo treatment mimicking 100.000 UI of cholecalciferol every 14 days for a maximum of 24 months or until conversion to full multiple sclerosis has occurred.
  Arms: Placebo
Other: Imaging — All patients are scheduled for MRI scans at baseline, 3 months, 12 months, 24 months, as well as upon conversion to full MS.
  Other Names: Cerebro-medullar MRI
Biological: Lumbar puncture — A baseline collection of cerebral spinal fluid may be required for certain patients (doctor's decision.)
Biological: Blood sampling — Blood sampling is required of all patients at baseline, 3 months, 6 months, 12 months, 18 months and 24 months, as well as upon conversion to MS.
Biological: Urine samples — Urine samples are required of all patients at baseline, 3 months, 6 months, 12 months, 18 months, 24 months, and upon conversion to MS.

SUMMARY:
The main objective of this study is to evaluate the efficacy and tolerance of 2 years of treatment with cholecalciferol (vitamin D3) in patients with a clinically isolated syndrome at high risk for MS (CIS).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. evaluate clinical efficacy: delay to conversion; number of relapses/episodes per year B. evaluate efficacy in terms of resonance imaging parameters (cerebral/spinal MRI) C. evaluate efficacy in terms of slowing the progression of disability as measured by EDSS score and subscores D. measure and assess cognitive abilities (PASAT) E. evaluate changes in quality of life (EQ5D questionnaires, SF36, and TLS-TLS-QoL10 COPING10), fatigue questionnaire (FSMC) and anxiety / depression questionnaire (HADS) F. evaluate treatment tolerance G. to correlate changes in clinical and imaging parameters with the evolution of serum levels of 25(OH)D2 and 25(OH)D3 H. establish a biobank of DNA and RNA from all patients in the study and conduct analyses of gene polymorphisms involved in the metabolism of vitamin D and the HLA system based on the increased levels of vitamin D after supplementation I. establish a biobank of CSF, plasma, blood cells, serum and RNA samples for patients in selected centers for research on prognostic biomarkers of conversion J. establish a biobank consisting of plasma tubes collected for the determination of 25-hydroxy-vitamin D K. Estimate the rate of discordance between the conversion decision made by the study neurologist and the result of the MRI re-interpretation performed at the end of the study as well as the proportion of patients identified a posteriori as as erroneously included according to the centralized reading.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 24 months of follow-up
* The patient has had a classic CIS with the past 90 days
* Reference cerebro-medullary MRI scheduled within the 90 days after the beginning of symptoms
* With MRI (cerebro ± medullary) showing demyelination according to spatial spread criteria by Swanton (2006):
* At least 1 lesion in at least 2 of the 4 following territories: (1) Peri-ventricular; (2) Juxta-cortical; (3) Sub-tentorial; (4) Medullary
* No other suspected pathology
* Vitamin D level in blood less than 100 nmol / l at the pre-inclusion visit
* Women of childbearing potential must use very effective contraception for the duration of the study. A very effective contraceptive method is defined as a method resulting in a low failure rate (that is to say less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, IUDs, sexual abstinence, or partner with a vasectomy.

Randomisation stratification criteria:

* The patient can also also meet the temporal dissemination criteria defined according to McDonald criteria 2010 (Polman et al., 2011), because this condition is currently not sufficient for prescribing a background treatment: Simultaneous presence of at least one asymptomatic lesion taking on contrast and at least one asymptomatic lesion not taking on contrast after injection of gadolinium

Exclusion Criteria:

* The patient is participating in another study (this criteria does not apply to the POLAR study (RCB 2011-A01269-32); patients included in this study may simultaneously participate in the POLAR study)
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Major medical or psychiatric illness that, according to the investigator, would result in the patient running an unnecessary risk or that could affect compliance with the study protocol
* Vitamin D insufficiency linked to currently active digestive or more general diseases (celiac disease, inflammatory bowel disease, intestinal bypass, short bowel syndrome, cirrhosis, nephrotic syndrome, hyperthyroidism, rickets, hypoparathyroidism, cancer, granulomatous diseases and lymphomas)
* Moderate or severe renal insufficiency (creatinine clearance less than 60 ml / min)
* Epilepsy not adequately controlled by treatment
* Any illness requiring chronic treatment with corticosteroids
* Patient with osteoporosis or history of osteopenia
* Pathology requiring calcium intakes greater than 1 gram per day
* Current or past history of hypercalcemia
* Medications that affect the metabolism of vitamin D other than corticosteroids; e.g. anticonvulsants [phenobarbital, primidone, phenytoin] rifampicin, isoniazid, ketoconazole, 5-FU and leucovorin, thiazide diuretics.
* Situations accompanied by increased vulnerability to hypercalcemia, e.g. arrhythmia or known heart disease, treatment with digitalis, and subjects with nephrolithiasis.
* Contraindications to vitamin D3 as mentioned in the documentation for UVEDOSE
* Known hypersensitivity to gadolinium and / or known inability to undergo an MRI (pacemaker, osteosynthesis material, intraocular metal splinter, etc ....).

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 316 (Actual)
Dates: Start 2013-07-16; Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Conversion to MS yes/no | 24 months
  Conversion to MS according to criteria described by McDonald (Polman et al 2005)

SECONDARY OUTCOMES:
Number of relapse episodes (number per year) | 24 months
number of new brain lesions found in FLAIR MRI or medullary lesions found in T2 MRI | 3 months
number of new brain lesions found in FLAIR MRI or medullary lesions found in T2 MRI | 12 months
number of new brain lesions found in FLAIR MRI or medullary lesions found in T2 MRI | 24 months
Number of new T1 lesions taking on Gadolinium highlighting | 3 months
  qualitative variable: 0, 1, or >1
Number of new T1 lesions taking on Gadolinium highlighting | 12 months
  qualitative variable: 0, 1, or >1
Number of new T1 lesions taking on Gadolinium highlighting | 24 months
  qualitative variable: 0, 1, or >1
Number of hyposignal T1 lesions (black holes) | 3 months
Number of hyposignal T1 lesions (black holes) | 12 months
Number of hyposignal T1 lesions (black holes) | 24 months
Lesional burden in mm^3 for each cerebral MRI | 3 months
Lesional burden in mm^3 for each cerebral MRI | 12 months
Lesional burden in mm^3 for each cerebral MRI | 24 months
Total number of Gadolinium highlighted lesions on T1 images | 3 months
  Exact number (semiautomatic measure)
Total number of Gadolinium highlighted lesions on T1 images | 12 months
  Exact number (semiautomatic measure)
Total number of Gadolinium highlighted lesions on T1 images | 24 months
  Exact number (semiautomatic measure)
Normalized cerebral volume (SIENAX) obtained from a T13D sequence | 3 months
  mm^3
Normalized cerebral volume (SIENAX) obtained from a T13D sequence | 12 months
  mm^3
Normalized cerebral volume (SIENAX) obtained from a T13D sequence | 24 months
  mm^3
Change in global cerebral volume (mm^3) | baseline versus 24 months
EDSS score, including all subscores | baseline
EDSS score, including all subscores | 3 months
EDSS score, including all subscores | 12 months
EDSS score, including all subscores | 24 months
EDSS score, including all subscores | after second MS episode (1st relapse)(maximum 24 months)
score for the PASAT 3 seconds section of the MSFC score | baseline
score for the PASAT 3 seconds section of the MSFC score | 3 months
score for the PASAT 3 seconds section of the MSFC score | 12 months
score for the PASAT 3 seconds section of the MSFC score | 24 months
score for the PASAT 3 seconds section of the MSFC score | after second MS episode (1st relapse)(maximum 24 months)
EQ5D questionnaire | baseline
EQ5D questionnaire | 3 months
EQ5D questionnaire | 12 months
EQ5D questionnaire | 24 months
SF36 questionnaire | baseline
SF36 questionnaire | 3 months
SF36 questionnaire | 12 months
SF36 questionnaire | 24 months
FSMC fatigue scale | baseline
FSMC fatigue scale | 3 months
FSMC fatigue scale | 12 months
FSMC fatigue scale | 24 months
TLS-QOL10 questionnaire | baseline
TLS-QOL10 questionnaire | 3 months
TLS-QOL10 questionnaire | 12 months
TLS-QOL10 questionnaire | 24 months
TLS-Coping10 questionnaire | baseline
TLS-Coping10 questionnaire | 3 months
TLS-Coping10 questionnaire | 12 months
TLS-Coping10 questionnaire | 24 months
HADS questionnaire | baseline
HADS questionnaire | 3 months
HADS questionnaire | 12 months
HADS questionnaire | 24 months
Presence/absence of adverse events | baseline
  Presence/absence of adverse events the severity of which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades I, II, III, IV, V.
Presence/absence of adverse events | 3 months
  Presence/absence of adverse events the severity of which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades I, II, III, IV, V.
Presence/absence of adverse events | 6 months
  Presence/absence of adverse events the severity of which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades I, II, III, IV, V.
Presence/absence of adverse events | 12 months
  Presence/absence of adverse events the severity of which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades I, II, III, IV, V.
Presence/absence of adverse events | 18 months
  Presence/absence of adverse events the severity of which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades I, II, III, IV, V.
Presence/absence of adverse events | 24 months
  Presence/absence of adverse events the severity of which will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades I, II, III, IV, V.
25(OH)D2+D3 serum level (nmol/l) | baseline
25(OH)D2+D3 serum level (nmol/l) | 3 months
25(OH)D2+D3 serum level (nmol/l) | 6 months
25(OH)D2+D3 serum level (nmol/l) | 12 months
25(OH)D2+D3 serum level (nmol/l) | 18 months
25(OH)D2+D3 serum level (nmol/l) | 24 months
25(OH)D2+D3 serum level (nmol/l) | upon conversion to MS (maximum 24 months)
Calciuria/creatinuria | baseline
Calciuria/creatinuria | 3 months
Calciuria/creatinuria | 6 months
Calciuria/creatinuria | 12 months
Calciuria/creatinuria | 18 months
Calciuria/creatinuria | 24 months
Calciuria/creatinuria | upon conversion to MS (maximum 24 months)
Delay until conversion to MS | 24 months
  The number of days that pass from the beginning of treatment to conversion to MS according to McDonald 2005 criteria (Polman et al 2005)

OTHER OUTCOMES:
DNA sample (blood sample) for biobank | baseline
Hemogram | baseline
Hemogram | 3 months
Hemogram | 6 months
Hemogram | 12 months
Hemogram | 18 months
Hemogram | 24 months
Hemogram | upon conversion to MS (maximum 24 months)
alanine amino transferase serum levels | baseline
alanine amino transferase serum levels | 3 months
alanine amino transferase serum levels | 6 months
alanine amino transferase serum levels | 12 months
alanine amino transferase serum levels | 18 months
alanine amino transferase serum levels | 24 months
alanine amino transferase serum levels | upon conversion to MS (maximum 24 months)
aspartate aminotransferase serum levels | baseline
aspartate aminotransferase serum levels | 3 months
aspartate aminotransferase serum levels | 6 months
aspartate aminotransferase serum levels | 12 months
aspartate aminotransferase serum levels | 18 months
aspartate aminotransferase serum levels | 24 months
aspartate aminotransferase serum levels | upon conversion to MS (maximum 24 months)
alkaline phosphatase serum levels | baseline
alkaline phosphatase serum levels | 3 months
alkaline phosphatase serum levels | 6 months
alkaline phosphatase serum levels | 12 months
alkaline phosphatase serum levels | 18 months
alkaline phosphatase serum levels | 24 months
alkaline phosphatase serum levels | upon conversion to MS (maximum 24 months)
serum calcium levels | baseline
serum calcium levels | 3 months
serum calcium levels | 6 months
serum calcium levels | 12 months
serum calcium levels | 18 months
serum calcium levels | 24 months
serum calcium levels | upon conversion to MS (maximum 24 months)
serum creatinine levels | baseline
serum creatinine levels | 3 months
serum creatinine levels | 6 months
serum creatinine levels | 12 months
serum creatinine levels | 18 months
serum creatinine levels | 24 months
serum creatinine levels | upon conversion to MS (maximum 24 months)
serum albumin levels | baseline
serum albumin levels | 3 months
serum albumin levels | 6 months
serum albumin levels | 12 months
serum albumin levels | 18 months
serum albumin levels | 24 months
serum albumin levels | upon conversion to MS (maximum 24 months)
serum urea levels | baseline
serum urea levels | 3 months
serum urea levels | 6 months
serum urea levels | 12 months
serum urea levels | 18 months
serum urea levels | 24 months
serum urea levels | upon conversion to MS (maximum 24 months)
serum bilirubin levels | baseline
serum bilirubin levels | 3 months
serum bilirubin levels | 6 months
serum bilirubin levels | 12 months
serum bilirubin levels | 18 months
serum bilirubin levels | 24 months
serum bilirubin levels | upon conversion to MS (maximum 24 months)
serum electrolyte panel | baseline
serum electrolyte panel | 3 months
serum electrolyte panel | 6 months
serum electrolyte panel | 12 months
serum electrolyte panel | 18 months
serum electrolyte panel | 24 months
serum electrolyte panel | upon conversion to MS (maximum 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvennot, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes; Eric Thouvenot, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (33):
- France (32):
  - CHU d'Amiens - Hôpital Nord, Amiens
  - CHU de Lyon - Hôpital Pierre Wertheimer, Bron
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHU de Clermont Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - CH Sud Francilien, Corbeil-Essonnes
  - Clinique des Cèdres - Capio, Cornebarrieu
  - CHU de Dijon, Dijon
  - CHU de Grenoble - Hôpital A Michallon, Grenoble
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Groupe Hospitalier de l'Institut Catholique de Lille, Lomme
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nancy - Hôpital Central, Nancy
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - CHU de Nice - Hôpital Pasteur, Nice
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - MAILLART Elisabeth - La Pitié Salpétrière, Paris
  - Fondation Ophtalmologique Adolphe Rothschild, Paris
  - APHP - Hôpital Saint-Antoine, Paris
  - CH de Pau, Pau
  - CH de Perpignan - Hôpital Saint Jean, Perpignan
  - CH de Cornouaille - Site Quimper - Hôpital Laennec, Quimper
  - CHU de Reims - Hôpital Maison Blanche, Reims
  - CHU de Rennes - Hôpital PontChaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CH de Poissy - Saint-Germain-en-Laye, Saint-Germain-en-Laye
  - CH de Saumur, Saumur
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg
  - CHRU de Toulouse - Hôpital Purpan, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours
  - CH de Versailles - Hôpital Mignot, Versailles
  - CH de Vichy - Jacques Larin, Vichy
- CHU de Martinique - Hôpital Pierre Zobda-Quitman, Fort-de-France, Martinique

REFERENCES:
- [Derived] Thouvenot E, Laplaud D, Lebrun-Frenay C, Derache N, Le Page E, Maillart E, Froment-Tilikete C, Castelnovo G, Casez O, Coustans M, Guennoc AM, Heinzlef O, Magy L, Nifle C, Ayrignac X, Fromont A, Gaillard N, Caucheteux N, Patry I, De Seze J, Deschamps R, Clavelou P, Biotti D, Edan G, Camu W, Agherbi H, Renard D, Demattei C, Fabbro-Peray P, Mura T, Rival M; D-Lay MS Investigators. High-Dose Vitamin D in Clinically Isolated Syndrome Typical of Multiple Sclerosis: The D-Lay MS Randomized Clinical Trial. JAMA. 2025 Apr 22;333(16):1413-1422. doi: 10.1001/jama.2025.1604. PMID 40063041

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT01817166/SAP_000.pdf